CLINICAL TRIAL: NCT07154472
Title: Upper Extremity Function in Individuals With Paraplegia: Relationships Between Endurance, Performance, and Symptoms
Brief Title: Upper Limb Function in Paraplegic Individuals: Exploring Endurance, Performance, and Symptoms
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, HÜSNA GÜZEL, lecturer, Hacettepe University
Other Study IDs: 24-282
Record Dates: First submitted 2025-08-08; First posted 2025-09-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Paraplegia; Endurance; Symptoms
Keywords: upper extremity; paraplegia; performance; symptoms
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Individuals with Paraplegia: The neurological impairment level of the individuals was assessed using the American Spinal Injury Association (ASIA) Classification, upper extremity endurance was evaluated with the 6-Minute Pegboard and Ring Test, upper extremity function was measured by the Purdue Pegboard Test, symptoms were assessed using the Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire, hand grip strength was measured with the Jamar hand dynamometer, functional independence was evaluated by the Functional Independence Measure (FIM), and physical activity level was assessed using the Physical Activity Scale for Individuals with Physical Disabilities.

SUMMARY:
Spinal cord injury (SCI) is a serious condition that causes physical, psychological, and social functional impairments. Paraplegia is characterized by the loss of motor and/or sensory function at the thoracic, lumbar, or sacral levels of the spinal cord, affecting the trunk, lower extremities, and pelvic organ functions. Functional independence and the ability to use a wheelchair are primary goals of rehabilitation. In paraplegia, the upper extremities are preserved; however, overuse often leads to shoulder and wrist pain and overuse injuries such as carpal tunnel syndrome. Pain is the most common symptom negatively impacting patients' quality of life. Additionally, findings such as decreased muscle strength, spasticity, atrophy, and joint limitations reduce functional performance. This study aims to investigate the relationships between upper extremity function (endurance and performance) and symptoms including pain, sensory loss, atrophy, joint limitations, and grip strength in individuals with paraplegia. Assessment methods used include the ASIA scale, 6-Minute Pegboard and Ring Test, Purdue Pegboard Test, DASH questionnaire, hand dynamometer, and Functional Independence Measure (FIM).

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a devastating condition that can cause physical, psychological, and social functional impairments. Paraplegia, a type of spinal cord injury, refers to the impairment or loss of motor and/or sensory functions of the thoracic, lumbar, or sacral spinal cord segments due to damage to neural structures within the spinal canal. Depending on the injury level, involvement of the trunk, lower extremities, and pelvic organs may occur.

Individuals with spinal cord injury need to have a good level of functional independence and the ability to use a wheelchair effectively in order to maintain their daily lives. Since individuals with SCI often rely heavily on wheelchairs during ambulation and daily activities, continuous load is placed on the bones, joints, and soft tissues of the upper extremities, which may lead to various upper limb problems.

Pain is the most common symptom affecting the quality of life in individuals with spinal cord injury. Additionally, shoulder pain, nerve neuropathies, motor and sensory loss, carpal tunnel syndrome, and muscle weakness can also be observed in these individuals.

Since paraplegic individuals must use a wheelchair, good upper extremity endurance is essential. However, there is a lack of studies in the literature assessing upper extremity endurance in this population. The performance of paraplegic individuals during daily activities is also important, yet no studies evaluating upper extremity performance in paraplegic individuals have been found. Our study is unique in that it aims to assess upper extremity endurance and performance in individuals with paraplegia.

In this study, the relationships between upper extremity function-endurance and performance-and symptoms such as pain, sensory loss, atrophy, joint restrictions, and grip strength associated with paraplegia were evaluated. The primary aim was to identify factors that hinder improvements in quality of life and independence by revealing the relationship between endurance, performance, and symptoms, and to provide data for rehabilitation programs to enhance the quality of life for these patients.

Thirty-two individuals with paraplegia participated in the study, which was conducted at Istinye University Physiotherapy and Rehabilitation Research and Application Center (İSÜFİZYOTEM). Neurological impairment was classified using the American Spinal Injury Association (ASIA) Impairment Scale. Upper extremity endurance was assessed with the 6-Minute Pegboard and Ring Test, upper extremity function with the Purdue Pegboard Test, symptoms with the Arm, Shoulder, and Hand Problems Questionnaire, hand grip strength with the Jamar dynamometer, functional independence with the Functional Independence Measure, and physical activity level with the Physical Activity Scale for Individuals with Physical Disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with paraplegia who use a wheelchair
* Classified as ASIA Impairment Scale grade A, B, or C
* Fully or partially dependent on a wheelchair
* Over 18 years of age
* Possessing sufficient upper extremity muscle strength required for wheelchair use

Exclusion Criteria:

* Individuals with spinal cord injuries outside the T6-T12 levels
* Presence of respiratory system diseases
* Presence of cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was conducted on individuals with paraplegia who applied to the İstinye University Physiotherapy and Rehabilitation Research and Application Center (İSÜFİZYOTEM).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
ASIA Scale | Day 1
  The most sensitive method for evaluating a patient with spinal cord injury is a standardized physical examination. The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), developed by the American Spinal Injury Association (ASIA) and also endorsed by the International Spinal Cord Society (ISCoS), has become the most widely used standardized clinical assessment and classification method worldwide in recent years.
6-Minute Pegboard and Ring Test (6PBRT) | Day 1
  Unsupported functional arm exercise capacity was assessed using the 6-Minute Pegboard and Ring Test (6PBRT). During the 6PBRT, patients sat in front of a board with two bars placed at individual shoulder height and width, with two additional bars positioned 20 cm above these, each holding ten rings. Participants were asked to practice by placing several rings before the test began. They were then instructed to move the rings as quickly as possible from the lower holes to the upper holes and back again for 6 minutes. Standardized encouragement was given every minute during the test. Systolic blood pressure (SBP), diastolic blood pressure (DBP) were measured using an aneroid sphygmomanometer (Erka, Bad Tölz, Germany), while heart rate (HR) and oxygen saturation (SpO2) were monitored with a pulse oximeter (Nonin Palmsat® 2500 series, Plymouth, MN, USA) both before and after the test. Perceived dyspnea, general fatigue, and arm fatigue were recorded using the Modified Borg Scale (mBS/0-10
PURDUE PEGBOARD TEST | Day 1
  After injuries, limitations in functional activities requiring fine motor skills that are commonly used in daily life have created the need to assess this function. The Purdue Pegboard Test, which evaluates fine motor skills, has become established in the healthcare field. It is suitable for assessing hand functions. The test consists of 5 subtests. One of these includes only a mathematical total score, while in the other 4 subtests, the individual actively performs tasks:
  Placing pins with the dominant hand (for 30 seconds) Placing pins with the non-dominant hand (for 30 seconds) Placing pins with both hands simultaneously (for 30 seconds) Mathematical total Placing pins, washers, and nuts (for 60 seconds) The test score is the total number of pins or pins, washers, and nuts placed at the end of the allotted time.
DASH Questionnaire | Day 1
  The Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) was developed in 1994 by the American Academy of Orthopaedic Surgeons (Hudak et al., 1996) to evaluate functional status and symptoms by focusing on physical function in upper extremity injuries.
  The DASH questionnaire consists of three sections. The first section contains 30 questions; 21 questions assess the patient's difficulty during daily living activities, 5 questions evaluate symptoms (pain, activity-related pain, tingling, stiffness, weakness), and the remaining 4 questions assess social function, work, sleep, and patient confidence.
  This first section determines the patient's Function/Symptom (DASH-FS) score. According to the DASH questionnaire results, a score between 0 and 100 is obtained for each section (0 = no disability, 100 = maximum disability).
Grip Strength | Day 1
  For the assessment of grip strength, the Jamar hand dynamometer (Fabrication Enterprises, New York, USA) was used, which is recommended by the American Society of Hand Therapists and is widely recognized in the literature for its high validity and reliability; therefore, it is considered the gold standard. Measurements were taken with the participant seated in an upright, supported position, with the elbow flexed at 90°, the arm adducted to the trunk, and the forearm in a neutral position. Assessments were performed three times for both the dominant and non-dominant hands, with a one-minute rest period between each measurement. The mean value of the three trials was recorded in kilograms-force (kgF) for both the affected and unaffected sides. In the interpretation of the results, the percentage of normative values based on age and gender was used.
Functional Independence Measure (FIM) | Day 1
  The Functional Independence Measure (FIM) is a widely used assessment tool developed to evaluate the level of functional independence in individuals with physical disabilities. It consists of 18 items, grouped under two major domains: motor (13 items) and cognitive (5 items). The motor domain includes self-care, sphincter control, mobility, and locomotion, while the cognitive domain evaluates communication and social cognition.
  Each item is scored on a 7-point ordinal scale, where:
  1 = total assistance required,
  7 = complete independence.
  The total FIM score ranges from 18 to 126, with higher scores indicating greater functional independence. FIM is commonly used in rehabilitation settings to track patient progress, evaluate treatment effectiveness, and plan discharge and follow-up care.
Assessment of Physical Activity Level: Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) | Day 1
  The Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) is a 13-item self-report questionnaire assessing daily activities, household tasks, and occupational roles over the past 7 days. It includes activities such as leisure-time exercise, sports, household chores, caregiving, and work-related tasks.
  Participants report the frequency (never to often) and duration (<1 hour to >4 hours/day) of each activity. The total score is calculated by multiplying the average time spent on each activity by its corresponding MET value. Item 1 is not scored and is intended for familiarization only.

CONTACTS AND LOCATIONS:
Overall Officials: Nurgül Dürüstkan Elbasi, asst. prof., Study Director — Istinye University; HÜSNA GÜZEL, PT,PhD (c), Study Chair — Istinye University; Berra Mina Eskili, student, Study Chair — Istinye University; Buse Deniz, STUDENT, Study Chair — Istinye University; OMER KACIRAL, STUDENT, Study Chair — Istinye University; HÜSNA GÜZEL, PT,PhD (c), Principal Investigator — Istinye University
Locations (1):
- Istinye University Physiotherapy and Rehabilitation Practice and Research Center, Istanbul, ZEYTINBURNU, Turkey (Türkiye)